CLINICAL TRIAL: NCT04298164
Title: Evaluating the Effectiveness of an Acceptance and Commitment Therapy-based Group Intervention for Parents of Children With a Diagnosis of Autism Spectrum Disorder Attending a Psychological Service
Brief Title: Evaluating the Effectiveness of an Acceptance and Commitment Therapy-based Group Intervention for Parents of Children With a Diagnosis of Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: START1
Record Dates: First submitted 2020-02-24; First posted 2020-03-06 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will generate a Unique Identifier Code which will be used to identify their data across each time point, but will mask their allocation until all of the data is entered and analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group that receives the intervention
  Interventions: Behavioral: START programme
- Control group (Active Comparator): Group that receives treatment as usual
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: START programme — Acceptance and Commitment Therapy based programme for parents of children with Autism
  Arms: Intervention group
Behavioral: Treatment as Usual — Treatment as usual in outpatient within outpatient psychology services
  Arms: Control group

SUMMARY:
This study is being conducted to look at whether a group programme designed for parents of children with a diagnosis of Autism is effective. The programme is called The START Programme ©- as it aims to provide a Supportive and Therapeutic environment to help parents gain Acceptance and reach Resolution so that they can Take action to live more consistently with their values. The programme was developed by two psychologists in Longford/Westmeath, Ireland, Dr. Michelle Howard and Kara McDermott in 2013, because they identified a lack of therapeutic support for such parents. The programme draws on research and theory from a branch of therapy called Acceptance and Commitment Therapy, as well as some other psychological techniques. Individuals who agree to participate in the research will be assigned at random to the intervention or to a treatment as usual control condition. They will be asked to fill out 4 questionnaires, on 3 different occasions, with a 7 week gap between the first time and second time, and a 3 month gap between the second and third time.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults over the age of 18 with the capacity to provide informed consent who are willing to take part in all aspects of the study
* They must have at least 1 child with a diagnosed autism spectrum disorder who is linked in with one of the psychology service sites involved in the study.
* They must not have completed the START programme before, or be concurrently attending another group based parental intervention.

Exclusion Criteria:

* Individuals who are under the age of 18, or who unable or unwilling to provide informed consent for all aspects of the study will be not included.
* Individuals who are receiving other current group based parental interventions will not be included.
* Couples may not attend the programme together, as outlined by the Psychologists who developed the programme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change in psychological flexibility | Measured before first session of programme (Week 1), at the final session of the programme (Week 7), and at 3 month follow up (12 Weeks after Week 7)
  Measured using the Comprehensive assessment of Acceptance and Commitment Therapy Processes (CompACT)

SECONDARY OUTCOMES:
Parenting stress | Measured before first session of programme (Week 1), at the final session of the programme (Week 7), and at 3 month follow up (12 Weeks after Week 7)
  Measured using The Autism Parenting Stress Index
Mental wellbeing | Measured before first session of programme (Week 1), at the final session of the programme (Week 7), and at 3 month follow up (12 Weeks after Week 7)
  Measured using The Warwick-Edinburgh Mental Wellbeing Scales (WEMWBS)
Parent relationship | Measured before first session of programme (Week 1), at the final session of the programme (Week 7), and at 3 month follow up (12 Weeks after Week 7)
  Parent Problem Checklist (PPC)

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - HSE Donegal, Donegal
  - HSE Longford/Westmeath, Longford

IPD SHARING:
Plan to Share IPD: No